CLINICAL TRIAL: NCT06472947
Title: Non-invasive Evaluation of Graft Condition in Adult Patients With Kidney Transplant Using Ultrasound Localization Microscopy and Multispectral Optoacoustic Tomography
Acronym: ESTIMATOR
Status: Recruiting | Type: Observational
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Principal Investigator, Ferdinand Knieling, Principal Investigator, Pediatric Translational Imaging Laboratory, University of Erlangen-Nürnberg Medical School
Other Study IDs: NTX_ULM_MSOT
Record Dates: First submitted 2024-06-18; First posted 2024-06-25 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Kidney Transplant; Kidney Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood and urine tests kidney tissue (biopsy)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient with kidney transplant: Included are adult (> 18 years) patients with kidney transplant where the indication for a kidney biopsy has been set during clinical routine
  Interventions: Device: ULM and MSOT

INTERVENTIONS:
Device: ULM and MSOT — transplanted kidney will be examined non-invasively with ULM and MSOT

SUMMARY:
In this study, the condition of the kidney transplant in adults is to be assessed non-invasively using Multispectral Optoacoustic Tomography and Ultrasound Localization Microscopy. New, non-invasive markers that allow conclusions to be drawn about the condition of the transplant should reduce the need for invasive diagnostic procedures in the future.

DETAILED DESCRIPTION:
In this study, the condition of the kidney transplant in adults is to be assessed non-invasively using multispectral multispectral optoacoustic tomography and ultrasound localization microscopy. Associated with common diseases such as arterial hypertension, diabetes mellitus and cardiovascular diseases, chronic renal failure is now a leading cause of death worldwide.

Around 10% of adults in Germany, but children are also affected. The terminal stage of renal insufficiency is defined by a glomerular filtration rate (GFR) which is only 15% of the normal rate and the need for renal replacement therapy in the form of dialysis or transplantation.

Not only the higher quality of life, but also the mortality rate make kidney transplantation the procedure of choice whenever possible.

After successful kidney transplantation, regular monitoring and evaluation of the organ transplant is of great importance to detect a rejection reaction as early as possible.

Among other things, this is done during an extensive annual examination. Not infrequently, and especially in the case of abnormalities in the laboratory diagnosis of blood and urine, a kidney biopsy is also necessary in order to assess the condition of the transplant in the best possible way.

As an invasive diagnostic procedure, the biopsy necessitates a stay in hospital, may result in side effects such as postoperative bleeding and represents a risk and an additional bruden for the patient.

MSOT has already been used to measure renal clearance and the biodistribution of fluorescent substances within the kidney, but new biomarkers have also been established in muscle and intestinal diseases and correlated with clinical scores. ULM has made the visualization of glomeruli, the smallest functional unit of the kidney, in living rats and humans and visualization of cerebral microvasculature in the human brain possible. In this study, the renal function in transplant patients will be evaluated as part of the annual examination and results from histology (biopsy), laboratory and ultrasound diagnostics will be correlated with data from MSOT and ULM imaging.

The investigators believe that MSOT can be used to gain important molecular insights into the condition of the transplant. With ULM the investigators want to analyze the microvascular architecture within glomerular renal corpuscles and identify changes in perfusion dynamics as morphological signs for transplant evaluation.

ELIGIBILITY:
Inclusion Criteria:

* kidney transplant
* indication for biopsy set in clinical routine
* minimum 18 years of age
* written consent

Exclusion Criteria:

* allergy against contrast agents/ SonoVue
* tatoos in examined areas
* contraindication against SonoVue
* pregnant women
* breast feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 10 patients with kidney transplant and indication for kidney biopsy
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2024-06-18 (Actual); Primary Completion 2025-06-18 (Estimated); Study Completion 2025-06-18 (Estimated)

PRIMARY OUTCOMES:
Visualization of microvascular architecture in the transplant kidney | Day1
  Using Ultrasound Localization Microscopy (ULM) for the non invasive visualization of microvasculature
Quantification of microvascular dynamics in the transplanted kidney | Day1
  Using Ultrasound Localization Microscopy (ULM) for the non invasive quantification of microvascular dynamics
MSOT in human kidney transplant | Day1
  Measuring MSOT signals (Signals for total/oxygenated/deoxygenated hemoglobin, lipid and collagen) in the human kidney transplant

SECONDARY OUTCOMES:
ULM visuals and histology | Day1
  ULM: Correlation of the vascular architecture of the transplant kidney visualized by ULM (e.g. number of segmented glomeruli) with histological parameters (e.g. Banff classification)
ULM visuals and laboratory results | Day1
  - ULM: Correlation of the vascular architecture of the transplant kidney visualized by ULM (e.g. number of segmented glomeruli) with laboratory chemical parameters (e.g. renal function parameters, inflammation parameters, immunological parameters)
ULM visuals and standard sonography | Day1
  - ULM: Correlation of the vascular architecture of the transplant kidney visualized by ULM (e.g. number of segmented glomeruli) with sonographic parameters (e.g. resistance index (RI), flow velocity)
ULM quantification and histology | Day1
  ULM: Correlation of parameters of quantified microvascular perfusion dynamics in the transplant kidney with histological parameters (e.g. Banff classification)
ULM quantification and laboratory results | Day1
  - ULM: Correlation of parameters of the quantified microvascular perfusion dynamics in the transplant kidney with laboratory chemical parameters (including renal function parameters, inflammation parameters)
MSOT: Hb and histology | Day1
  MSOT: Correlation of the signal determined with MSOT for total/oxygenated/deoxygenated
MSOT: hb and laboratory results | Day1
  - MSOT: Correlation of the signal for total/oxygenated/deoxygenated hemoglobin with laboratory chemical parameters
MSOT hb and sonography | Day1
  - MSOT: Correlation of the signal for total/oxygenated/deoxygenated hemoglobin determined with MSOT with sonographic parameters
MSOT hb and histology | Day1
  - MSOT: Correlation of the signal for total/oxygenated/deoxygenated hemoglobin with with histological parameters
MSOT Lipid and laboratory results | Day1
  - MSOT: Correlation of the signal for lipid determined with MSOT with laboratory chemical parameters
MSOT Lipid and sonographic results | Day1
  MSOT: Correlation of the signal for lipid determined with MSOT with sonographic parameters parameters
MSOT lipid and histology | Day1
  MSOT: Correlation of the signal for lipid determined with MSOT with histological parameters
MSOT collagen and sonography | Day1
  - MSOT: Correlation of the signal for collagen determined with MSOT with sonographic parameters
MSOT collagen and histology | Day1
  MSOT: Correlation of the signal for collagen determined with MSOT with histological parameters
MSOT collagen and laboratory results | Day1
  - MSOT: Correlation of the signal for collagen determined with MSOT with laboratory chemical parameters
ULM quantification and sonography | Day1
  Correlation of parameters of the quantified microvascular perfusion dynamics in the transplant kidney with sonography in transplanted kidney

CONTACTS AND LOCATIONS:
Overall Officials: Ferdinand Knieling, PD Dr. Dr., Principal Investigator — FAU Erlangen-Nuremberg
Locations (1):
- Department of Pediatrics and Adolescent Medicine, Erlangen, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No